CLINICAL TRIAL: NCT01993550
Title: Telephone Symptom Management for Advanced Lung Cancer Patients and Caregivers
Brief Title: Telephone Support Program for Lung Cancer Patients and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other); American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1K07CA168883-01A1 (NIH); 1K07CA168883-01A1 (NIH)
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; family caregiving; behavioral intervention; counseling; symptom management
MeSH Terms: conditions — Lung Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone counseling (Experimental): Telephone counseling to enhance symptom management and reduce distress
  Interventions: Behavioral: Telephone counseling
- Education (Active Comparator): Overview of resources for psychosocial support and health information
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Telephone counseling
  Arms: Telephone counseling
Behavioral: Education
  Arms: Education

SUMMARY:
The goal of this project is to examine the physical and psychological health benefits of a novel, telephone-delivered symptom management intervention for advanced lung cancer patients and their family caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lung cancer
* Must be able to speak and read English

Exclusion Criteria:

* No working phone service
* Does not have a family caregiver

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-8 | baseline, 2 and 6 weeks post-intervention
Change in Generalized Anxiety Disorder 7-item scale | baseline, 2 and 6 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E. Mosher, Ph.D., Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winger JG, Rand KL, Hanna N, Jalal SI, Einhorn LH, Birdas TJ, Ceppa DP, Kesler KA, Champion VL, Mosher CE. Coping Skills Practice and Symptom Change: A Secondary Analysis of a Pilot Telephone Symptom Management Intervention for Lung Cancer Patients and Their Family Caregivers. J Pain Symptom Manage. 2018 May;55(5):1341-1349.e4. doi: 10.1016/j.jpainsymman.2018.01.005. Epub 2018 Jan 31. PMID 29366911